CLINICAL TRIAL: NCT05894070
Title: The Voice as a Tool to Detect Recurrence of Laryngeal and Hypopharyngeal Cancer (VoiceDetect) - a Feasibility Study
Brief Title: The Voice as a Tool to Detect Recurrence of Laryngeal and Hypopharyngeal Cancer
Acronym: VoiceDetect
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-00838
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Laryngeal Cancer; Hypopharyngeal Cancer
MeSH Terms: conditions — Laryngeal Neoplasms; Hypopharyngeal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Voice recording, ENT (Ear, Nose and Throat) examination including transnasal fiberendoscopy, and VHI-30-questionnaire — The following speech samples will be recorded from the study participants:
  * Standardized, phonetically balanced text
  * Sustained, modulated production of five vowels
  * Picture description
  * Diadochokinetic exercise.
  Before starting speech recording, the participant fills in a questionnaire consisting of:
  * Health barometer
  * Self-rating in terms of stress/fatigue/emotional status.
  An Ear, Nose and Throat examination incl. transnasal fiberendoscopy is performed at each visit. The investigators will assess the vocal folds/aryepiglottic folds for the presence of paralysis or reduced mobility, as well as the presence of scar/synechia, edema, erythro-/leukoplakia, or a cancer-suspicious lesion/mass in the larynx/hypopharynx or a chondroradionecrosis in the larynx.
  Additionally, it will be assessed, if a tracheotomy canula or a nasogastric tube is in place or was used since the last visit.
  Furthermore, the investigators will ask the patients to fill out the VHI-30.

SUMMARY:
The investigators will obtain three-monthly voice recordings and fiberendoscopic examinations of the larynx/hypopharynx for a minimal period of 6 months from all laryngeal/hypopharyngeal squamous cell carcinoma (LSCC/HPSCC) patients, who have successfully completed curative primary treatment, except those who underwent total laryngectomy. Furthermore, the investigators will ask the patients to fill out the voice handicap index-30 questionnaire (VHI-30) during each study visit. The VHI-30 allows to make a subjective assessment of the patients' own vocal problem. The primary objective is to assess the feasibility and compliance of longterm regular voice monitoring in LSCC and HPSCC follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically proven carcinoma in-situ or invasive LSCC or HPSCC (in non-surgically treated carcinoma: clinical/radiologic stage I-IV (excluding M1) according to the Union for International Cancer Control (UICC) / Tumor (T), Nodes (N), and Metastases (M) (TNM) 8th ed.; in surgically treated carcinoma: pathological stage I-IV (excluding M1) according to the UICC / TNM 8th ed.).
2. ≥ 18 years of age.
3. Treatment with curative intent, regardless of treatment modality (mono- or multimodal).

   Remark: Patients with synchronous (larynx and hypopharynx included) or metachronous (before/after the diagnosis of LSCC/HPSCC) non-laryngeal/-hypopharyngeal malignant non-metastatic tumors, with clinically confirmed complete remission 6 months after treatment and life expectancy of at least 6 months are eligible. Patients with surgically treated Tis-2 N0 M0 squamous cell carcinoma and/or basal cell carcinoma of the skin and/or other surgically treated non-head and neck Tis are eligible, although the treatment was within the 6 months before enrolment.
4. Clinical confirmation of complete remission of LSCC or HPSCC through Ear, Nose and Throat (ENT) examination, including fiberendoscopy of the pharynx and larynx, at the time of enrolment, during the period of eligibility (6 to 30 months after treatment).

   Remark: Patients with synchronous (larynx and hypopharynx included) or metachronous (before/after the diagnosis of LSCC/HPSCC) non-laryngeal/-hypopharyngeal malignant non-metastatic tumors, with clinically confirmed complete remission 6 months after treatment and life expectancy of at least 6 months are eligible. Patients with surgically treated Tis-2 N0 M0 squamous cell carcinoma and/or basal cell carcinoma of the skin and/or other surgically treated non-head and neck Tis are eligible, although the treatment was within the 6 months before enrolment.
5. Informed consent as documented by signature.

Exclusion Criteria:

1. Total laryngectomy as primary therapy.
2. Any local, regional, and systemic laryngeal or hypopharyngeal cancer persistence/progression, or recurrence before enrolment.

   Excepted: Patients with synchronous laryngeal/hypopharyngeal malignant non-metastatic tumors, with clinically confirmed complete remission 6 months after treatment and life expectancy of at least 6 months are eligible.
3. Any local, regional, and systemic tumor persistence/progression, or recurrence of synchronous (larynx and hypopharynx included) or metachronous (before/after the diagnosis of LSCC/HPSCC) non-laryngeal/-hypopharyngeal malignant tumors within 6 months before enrolment.

   Excepted: Patients with surgically treated progredient or recurrent locally defined Tis-2 N0 M0 squamous cell carcinoma and/or basal cell carcinoma of the skin and/or non-head and neck progredient or recurrent Tis.
4. Any previously treated LSCC/HPSCC or treated second primary malignancies of the larynx or hypopharynx before the diagnosis and treatment of the investigated LSCC/HPSCC (= index tumor).
5. Presence of any medical, psychological, familial, sociological, or geographical conditions expected to potentially hamper the compliance with the study protocol.
6. Inability to follow procedures (e.g., inability to read) or insufficient knowledge of any project language (German and French).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The anticipated study population are patients with LSCC and HPSCC who have successfully completed curative, organ-preserving primary treatment and did not show tumor persistence, recurrence, or second primary malignancy prior to the recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Patients' compliance with scheduled 3-monthly endoscopic exam, voice recordings, and filling out of questionnaire | 3-21 months
  The number of completed visits/exams out of all scheduled visits/exams.
Recruitment rate | 0-21 months
  Recruitment rate (number of enrolled participants per year).

SECONDARY OUTCOMES:
Subjective changes in voice | 0-21 months
  Subjective changes in voice assessed by the voice handicap index-30 (VHI-30).
Objective changes in voice 1 | 0-21 months
  Changes in Roughness - Breathiness - Hoarseness (RBH).
Objective changes in voice 2 | 0-21 months
  Changes in Jitter and Shimmer (JS).
Objective changes in voice 3 | 0-21 months
  Changes in Glottal-to-Noise Excitation Ratio (GNE).
Objective changes in voice 4 | 0-21 months
  Changes in Singing Power Ratio (SPR).
Recurrences of the index tumor | 0-21 months
  Number/Percentage of patients with biopsy-proven local, regional, and/or systemic recurrences of the initially treated LSCC/HPSCC.
  Note: In special scenarios such as co-morbidities, patient's rejection or other medical conditions, a biopsy can be omitted if there is a consensus for a recurrence at the multidisciplinary tumor board based on the clinical and/or radiologic findings.
Recurrences in other localizations | 0-21 months
  Number/Percentage of patients with biopsy-proven local, regional, and/or systemic recurrences in other localizations.
  Note: In special scenarios such as co-morbidities, patient's rejection or other medical conditions, a biopsy can be omitted if there is a consensus for a recurrence at the multidisciplinary tumor board based on the clinical and/or radiologic findings.
Second primary malignancies in the larynx/hypopharynx | 0-21 months
  Number/Percentage of patients with biopsy-proven local, regional, and/or systemic second primary malignancy in the larynx/hypopharynx.
  Note: In special scenarios such as co-morbidities, patient's rejection or other medical conditions, a biopsy can be omitted if there is a consensus for a second primary malignancy at the multidisciplinary tumor board based on the clinical and/or radiologic findings.
Second primary malignancies in other localizations | 0-21 months
  Number/Percentage of patients with biopsy-proven local, regional, and/or systemic second primary malignancy in other localizations.
  Note: In special scenarios such as co-morbidities, patient's rejection or other medical conditions, a biopsy can be omitted if there is a consensus for a second primary malignancy at the multidisciplinary tumor board based on the clinical and/or radiologic findings.
Composite of clinical events | 0-21 months
  Composite endpoint: Number/Percentage of patients with laryngeal/hypopharyngeal recurrence, second primary malignancy, edema, scar/synechia, erythro-/leukoplakia, laryngeal chondroradionecrosis and hypomobility/ paralysis determined by fiber-endoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Roland Giger, Prof., Principal Investigator — Inselspital, Bern University Hospital
Locations (2):
- Switzerland (2):
  - Department of Oto-Rhino-Laryngology, Head and Neck Surgery, Inselspital, Bern University Hospital, Bern
  - Department of Oto-Rhino-Larnygology, Head and Neck Surgery, University Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No